CLINICAL TRIAL: NCT05171023
Title: Application of ROTEM Technology in Aortic Surgery Under Cardiopulmonary Bypass and Circulatory Arrest
Brief Title: Application of ROTEM Technology in Aortic Surgery
Status: Completed | Type: Observational
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Aleksandr Eremenko, Clinical Professor, Petrovsky National Research Centre of Surgery
Other Study IDs: 20210916-11
Record Dates: First submitted 2021-11-16; First posted 2021-12-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Aortic Surgery; Coagulation Management
Keywords: ROTEM; coagulation tests; coagulation disorders; aortic surgery
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ROTEM and standard coagulation tests — ROTEM and standard coagulation tests assessment

SUMMARY:
Comparison of the diagnostic capabilities of rotational thromboelastometry (ROTEM) and standard coagulogram in the detection of disorder and correction of the hemostasis system in the perioperative period in patients who underwent surgical intervention on the aorta under cardiopulmonary bypass and or circulatory arrest.

DETAILED DESCRIPTION:
The patient is monitored in the intensive care unit according to the following scheme: ROTEM (NATEM, INTEM, EXTEM, FIBTEM; with high clotting time (CT) values in INTEM - HEPTEM is done) and a coagulogram (activated coagulation time (ACT), activated partial thromboplastin time (APTT), prothrombin time (PT), thrombin time (TT), fibrinogen, antithrombin III, platelet aggregation) are done on admission and after 6 hours - with a smooth course of the perioperative period. If it is necessary or the development of disorders in the form of bleeding or thrombosis that require correction, ROTEM and a coagulogram are done, treatment is carried out, and after elimination of the causes, ROTEM and a coagulogram are examined in dynamics to assess the effectiveness of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 80 years.
* Patients after surgical interventions on the aorta with cardiopulmonary bypass and/or circulatory arrest (operations on the ascending aorta, aortic arch and thoracoabdominal aorta).

Exclusion Criteria:

* Patients with other cardiac surgery, including isolated endovascular interventions on the aorta.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after surgical interventions on the aorta with cardiopulmonary bypass and/or circulatory arrest.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
The coagulation index | an average of during the first day after surgery
  Сhanges of the coagulation index
Activated coagulation time | an average of during the first day after surgery
  Сhanges of the activated coagulation time

SECONDARY OUTCOMES:
Percentage of repeated operations | an average of 24 hours after surgery
  Percentage of repeated operations
Percentage of multiple organ failure | an average of 24 hours after surgery
  Percentage of multiple organ failure
Percentage of serious infectious complication | an average of 24 hours after surgery
  Percentage of serious infectious complication

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Eremenko, MD, Study Director — Petrovsky National Research Centre of Surgery
Locations (1):
- Petrovsky National Research Centre of Surgery, Moscow, Russia